CLINICAL TRIAL: NCT02741011
Title: Computed Tomographic Assessment of the Maxillofacial Region of Mentally Handicapped or Uncooperative Patients Under Intravenous Sedation
Brief Title: Radiological Examination of the Mentally Handicapped Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tokat Gaziosmanpasa University (Other)
Responsible Party: Principal Investigator, Emrah Soylu, Asistan Professor, Tokat Gaziosmanpasa University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: ES-Tez01
Record Dates: First submitted 2016-02-24; First posted 2016-04-18 (Estimated); Last update posted 2016-04-18 (Estimated); Status verified 2016-04

CONDITIONS: Profound Mental Retardation
Keywords: Cone-Beam Computed Tomography; Mentally Handicapped
MeSH Terms: conditions — Intellectual Disability | interventions — X-Rays

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Radiological imaging (Other): Mentally handicapped patients underwent sedation anesthesia with IV Propofol and then tomographic images were obtained with NewTom 5G. Orthopantomographies (OPGs) were obtained by processing the raw images and radiological examination of the patients were performed on OPGs.
  Interventions: Other: Radiological examination

INTERVENTIONS:
Other: Radiological examination — During the period of two years, mentally handicapped patients were enrolled in this study. First a radiological examination was performed under sedation anesthesia and then an oral examination was performed when patient underwent general anesthesia for dental treatments. Oral and radiological examinations were compared with each other and also with treatment results to define the necessity of the radiological examination of mentally handicapped patients.

SUMMARY:
Aim of this study is to evaluate the necessity of the radiological examinations of mentally handicapped or uncooperative patients.

DETAILED DESCRIPTION:
Dental radiography has become an indispensable part of routine dental examination with the help of the technological development of radiological devices. However, medical procedures like dental treatment and medical imaging (magnetic resonance imaging-MRI, computed tomography-CT, orthopantomography- OPG, etc.) that require cooperation are usually hard to apply to mentally handicapped (MHP) or uncooperative patients (UCP). Treatments that will be done without radiological examination can be missing or incorrect.

ELIGIBILITY:
Inclusion Criteria:

1. Mentally Handicapped patients that radiological examination cannot performed
2. Suitable for IV sedation

Exclusion Criteria:

1. Healthy Patients
2. Patients in which the radiological examination performed

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2012-02; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Comparison of the radiological and oral examinations in mentally handicapped patients | 2 years
  Radiological images of the mentally handicapped patients obtained under sedation anesthesia with cone beam dental tomography. Radiological examination were performed on tomograpic images and indications (tooth filling, root canal treatment, extraction) were noted. Same procedure was performed for oral examination and indications were compared.

IPD SHARING:
Plan to Share IPD: No